CLINICAL TRIAL: NCT05709873
Title: Behavioral Treatment of Narcolepsy-Related Nightmares
Brief Title: Narcolepsy Nightmare Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU00218129
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Narcolepsy; Narcolepsy Type 1; Narcolepsy With Cataplexy; Narcolepsy Type 2; Narcolepsy Without Cataplexy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Imagery rehearsal therapy (IRT) (Experimental): Participants randomized to this group will receive 7 sessions of IRT.
  Interventions: Behavioral: Imagery rehearsal therapy
- Imagery rehearsal therapy and targeted dream control (IRT+TDC) (Experimental): Participants randomized to this group will receive 7 sessions of IRT+TDC.
  Interventions: Behavioral: Imagery rehearsal therapy; Behavioral: Targeted dream control

INTERVENTIONS:
Behavioral: Imagery rehearsal therapy — Therapy to reduce nightmares, delivered via videoconference sessions
  Other Names: IRT
Behavioral: Targeted dream control — Therapy to reduce nightmares, delivered in videoconference sessions and lab session. Lab session will involve a sleep study during a daytime nap.
  Other Names: TDC
  Arms: Imagery rehearsal therapy and targeted dream control (IRT+TDC)

SUMMARY:
The goal of this clinical trial is to test two behavioral treatments for nightmares in adults with narcolepsy. The main questions it aims to answer are:

* Is imagery rehearsal therapy (IRT) effective for narcolepsy-related nightmares?
* Does adding targeted dream control (TDC) to IRT make it more effective?

Participants will be randomized to one of two treatment groups and will be asked to:

* Complete a daily log of sleep symptoms for up to 13 weeks.
* Attend 7 sessions of treatment.
* Complete questionnaires before and after treatment.
* Go to the research lab in Evanston, IL to complete a sleep study during a daytime nap (Chicago area residents only).

ELIGIBILITY:
Inclusion Criteria (all participants):

* Diagnosis of narcolepsy
* Age 18 or older
* Speak English
* Live in the United States
* Receiving standard medical care for narcolepsy
* Sleep and psychiatric medications stable for at least 3 months
* Nightmare frequency of ≥3 times per week
* Nightmare Disorder Index score indicates probable nightmare disorder

Inclusion Criteria (Chicago area participants):

* Able to attend a study appointment in Evanston, IL
* Able and willing to not take wake-promoting medications on day of lab visit

Exclusion Criteria:

* History of a neurological disorder that might alter EEG
* Currently engaged in sleep- or trauma-focused psychotherapy
* Previous behavioral treatment for nightmares
* Medical, psychiatric, or cognitive condition which would interfere with ability to engage in the treatment
* Untreated sleep apnea (AHI ≥ 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Daily diary | Duration of study (11-13 weeks)
  Nightmare severity/frequency

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mundt, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States